CLINICAL TRIAL: NCT06087523
Title: Prevalence of Pulmonary Diseases Among Patients With Systemic Lupus Erythematosus, a Population-Based Cross-Sectional Study
Brief Title: Pulmonary Disease Among Patients With Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Vejle Hospital (Other); Sonderborg Hospital (Other Government)
Responsible Party: Principal Investigator, Anne Voss, MD, PhD, Professor, Odense University Hospital
Other Study IDs: OP_1858
Record Dates: First submitted 2023-09-08; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Lupus Erythematosus, Systemic; Pulmonary Disease
Keywords: Lupus Erythematosus, Systemic; Pulmonary Disease; Ultrasonography; Autoantibodies; Patient Reported Outcome Measures; Respiratory Function Tests; Tomography, Spiral Computed
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lung Diseases | interventions — Respiratory Physiological Phenomena; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples, serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multidisciplinary discussion — Multidisciplinary discussion: Participants will be diagnosed and categorized in regards of pulmonary disease on basis of medical record, PFT, HRCT, and questionnaires.
  PFT: Participants will undergo body plethysmography (with diffusion) and six-minute walk test.
  Analysis of circulating biomarkers: We will store glasses with serum and glasses with plasma and analyse them for circulating biomarker.
  Questionnaires: Participants will complete Danish versions of three questionnaires.
  * Saint George's Respiratory Questionnaire Interstitial Pulmonary Fibrosis
  * Systemic Lupus Activity Questionnaire
  * Lupus Impact Tracker
  Review of medical record and clinical investigation with focus on SLE and pulmonary disease.
  Thoracic and diaphragmatic ultrasound: The participants will undergo a 14 zone protocol, and be evaluated for b-lines and pleural thickening/irregularities. Diaphragm function will be evaluated according to the M-mode method, area method, and for thickening.
  Other Names: Thoracic and diaphragmatic ultrasound; High resolution CT scan of thorax (HRCT); Pulmonary function testing (PFT); Analysis of circulating biomarkers; Questionnaires (PROMs); Review of medical record.; Clinical investigation

SUMMARY:
Pulmonary diseases are common among patients with Systemic Lupus Erythematosus (SLE) and associated with a significantly increased morbidity, mortality, and lower self-reported health related quality of life.

The investigators aim to diagnose and categorise SLE patients in regards of pulmonary disease and introduce alternative diagnostic tools.

The investigators will perform a cross-sectional study of a population-based study population of SLE patients. The participants will undergo review of medical record, a clinical assessment, body plethysmography, six-minute walk test, high-resolution computed tomography of the thorax (HRCT), thoracic and diaphragmatic ultrasound, blood sampling with analysis of autoantibodies, and three questionnaires. After the investigations, pulmonary diseases among the participants will be diagnosed at a multidisciplinary discussion by a specialised pulmonologist with contribution from a rheumatologist and a radiologist.

The investigators believe that the study will increase the understanding of pulmonary diseases among SLE patients, which could improve overall disease management. The investigators will introduce new alternative diagnostic tools, that could ease diagnosing pulmonary disease among SLE.

DETAILED DESCRIPTION:
Background Pulmonary diseases are common among patients with Systemic Lupus Erythematosus (SLE) and cover a variety of manifestations including pleuritis and interstitial lung disease. Pulmonary diseases among SLE patients are associated with an increased morbidity, mortality, and lower self-reported health related quality of life.

Objective The primary objective of the study is to diagnose and categorise a population-based study population of SLE patients in regards of pulmonary diseases. The secondary objective of the study is to introduce alternative diagnostic tools to diagnose pulmonary disease among SLE patients, including thoracic ultrasound and circulating biomarkers.

Methods and Analysis The study will be reported according to the STROBE guidelines. The investigators will perform a cross-sectional study of a population-based study population of SLE patients. The participants will undergo review of medical record, a clinical assessment, body plethysmography, six-minute walk test, HRCT, thoracic and diaphragmatic ultrasound, blood sampling with analysis of autoantibodies, and three questionnaires translated to Danish - Saint George's Respiratory Questionnaire, Systemic Lupus Activity Questionnaire, and Lupus Impact Tracker. After the investigations, pulmonary diseases among the participants will be diagnosed at a multidisciplinary discussion by a specialised pulmonologist with contribution from a rheumatologist and a radiologist. The results will be blinded to the investigators except for Henrik Zachar Langkilde who will have access to results (except for the MDD diagnose) while the investigations are performed, and before the unblinding a statistical analyse plan will be reported. At the second of October 22 participants have had a visit.

Discussion Pulmonary diseases among SLE patients are common and of importance to the patients, but an area not studied as extensively as other disease manifestations. The investigators believe that this study will increase the understanding of pulmonary disease among SLE patients, which could improve overall disease management for the patients. The investigators hope that the alternative diagnostic tools introduced will ease to diagnose pulmonary disease among SLE patients. The study is approved by the Committees on Health Research Ethics and an umbrella organisation under the Danish Data Protection agency. The project, the protocol and the study design are discussed with two SLE patient partners, and the patient partners suggestions have been incorperated in the project.

ELIGIBILITY:
Inclusion Criteria:

* Followed at a Department of Rheumatology in Region Southern Denmark.
* Living in Region Southern Denmark.
* Diagnosed with Systemic Lupus Erythematosus.
* Fulfil the 2019 European League Against Rheumatism / American College of Rheumatology classification criteria.
* Speak and understand spoken and written Danish

Exclusion Criteria:

* Participants not having their native lungs
* Not participating in visit day, without a valid reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Systemic Lupus Erythematosus, in Region Southern Denmark (approximately 300 individuals)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of pulmonary diseases | From visit date to diagnose is noted, up to six weeks
  Participants will be diagnosed and categorised in regards of pulmonary disease at a multidisciplinary discussion the investigators will note following pulmonary diseases:
  * Pleural disease
  * Airway disease
  * ILD
  * Shrinking lung syndrome
  * Vascular Disease
  * Malignancy
  The diagnosis will be associated to PFT, PROMs, and HRCT.
  PFT:
  * Body plethysmography
  * Lung diffusion testing
  * Six-minutes walk test.
  HRCT, note presence of
  * ILD
  * Airway disease
  * Pleural disease
  * Vascular disease
  PROMs:
  * Saint George's Respiratory Questionnaire Interstitial Pulmonary Fibrosis (SGRQi)
  * Systemic Lupus Activity Questionnaire (SLAQ)
  * Lupus Impact Tracker (LIT)

SECONDARY OUTCOMES:
Ability of alternative diagnostic tools for diagnosis of pulmonary disease in patients with SLE as compared to gold standard | Thoracic ultrasound, diaphragmatic ultrasound, clinical investigations of patients, PFT, HRCT and PROMs are noted with a month after the visit.
  Results from thoracic ultrasound, diaphragmatic ultrasound, analysis of circulating biomarkers, clinical investigation of patients, and medical record will be associated to the diagnose from the multidisciplinary discussion, PFT, HRCT, and PROMs, as noted above.
  Thoracic ultrasound
  * Number of b-lines
  * Pleural irregularities
  Diaphragmatic ultrasound
  * M-mode method
  * Area method
  * Diaphragmatic thickness
  Circulating biomarkers. The biomarkers are not decided yet.
  Review of medical record, the investigators will note. - Prior diagnoses, chest immaging, blood and urine samples.
  Clinical investigation and medical interview, the investigator will score according to:
  * SLEDAI-2k
  * PGA
  * SLICC/ACR DI
  * LLDAS
  * DORIS
  and
  - note changes of the extremities and auscultate the lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Voss, MD, PhD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Region Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No